CLINICAL TRIAL: NCT00653991
Title: SOLVE IT: Real Risk Reduction for MSM
Brief Title: The SOLVE-IT National Randomized Trial
Acronym: SOLVE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lynn Miller, Study Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH082671 (NIH); R01MH082671 (NIH); DAHBR 9A-ASPQ (Other: NIMH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: HIV Infections
Keywords: HIV/AIDS Prevention; Men Who Have Sex With Men (MSM); Risky Sexual Behavior; Socially Optimized Learning in a Virtual Environment (SOLVE); HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOLVE-IT (Experimental): Participants will receive the intervention SOLVE-IT. The SOLVE-IT intervention is a videogame designed to optimize self-regulation, reduce shame, and reduce risky choices for young men who have sex with men (YMSM).
  Interventions: Behavioral: SOLVE-IT
- Waitlist Control (Active Comparator): Participants will receive the intervention, SOLVE-IT, a video game designed to optimize self-regulation reduce shame, and reduce risky sexual choices for YMSM, after a 6-month waitlist period.
  Interventions: Behavioral: SOLVE-IT

INTERVENTIONS:
Behavioral: SOLVE-IT — SOLVE-IT, a video game using computer-generated virtual agents, is the next generation of interactive media aimed at reducing risky sex among young MSM. Participants will interact in a virtual environment that focuses upon HIV prevention in a dating context.
  Other Names: Socially Optimized Learning in Virtual Environments

SUMMARY:
This study will evaluate the effectiveness of an interactive virtual environment computer game in reducing risky sexual behaviors among men who have sex with men.

DETAILED DESCRIPTION:
HIV and sexually transmitted diseases (STDs) are a major public health concern worldwide. Although prevalent across all groups of people, HIV/STDs have had a remarkable effect on men who have sex with men (MSM), who accounted for 71% of all HIV infections among American males in 2005. After years of decline, the number of HIV diagnoses appears to have increased for MSM, especially within the black MSM population. Thus, new approaches geared for HIV prevention and education and built on past HIV prevention methods are needed. New technologies, such as interactive computer games, delivered in a modern and appealing manner may gain or recapture the attention of MSM who have disregarded more traditional HIV prevention and educational services. Socially Optimized Learning in a Virtual Environment (SOLVE)-IT is an interactive virtual environment computer game, designed specifically for MSMs, that simulates the emotional, interpersonal, and contextual narrative of an actual sexual encounter and provides challenging decision-making opportunities. By promoting development of self-regulatory and behavioral skills, SOLVE-IT may be an effective approach to reduce sexual risk behaviors. This study will evaluate the effectiveness of SOLVE-IT in reducing risky sexual behaviors among MSM.

Participation in this study will last 6 months from the beginning of treatment. All participants will first undergo baseline assessments that will include questionnaires about sexual behavior, drug use, health history, feelings, and beliefs. Participants will then be assigned randomly to receive SOLVE-IT immediately or after a 6-month waitlist period. SOLVE-IT will include two 1-hour sessions conducted on a computer over the Internet, occurring at baseline and 6 months later. During sessions, participants will play an interactive computer game that presents dating or sexual scenarios and allows participants to choose how the scenarios unfold. Participants will repeat baseline questionnaires at Months 3 and 6 of follow-up. Participants in the waitlist group will be offered to receive SOLVE-IT after completion of the Month 6 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Latino, black, or Caucasian
* Men who have sex with men
* Not HIV infected
* Engaged in unprotected anal sex at least twice in the 90 days before study entry with a nonprimary male partner
* Has broadband access during course of study
* Lives in United States
* Biological male

Exclusion Criteria:

* History of nonprescription drug injection use
* Has participated in SOLVE-IT at any phase

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2020 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn C. Miller, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California (University Village), Los Angeles, California, United States

REFERENCES:
- [Background] Read SJ, Miller, LC, Appleby PR, Nwosu ME, Reynaldo S, Lauren A, Putcha A. Socially optimized learning in a virtual environment: Reducing risky sexual behavior among men who have sex with men. Human Communication Research 32(1):1-34, 2006.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Allocation 1284 SOLVE-IT (Met exclusion: 573 incomplete baseline; 257 didn't play game; 10 technical glitch)
  2. Allocation 736 Control (Met exclusion: 202 didn't complete baseline; 43 had technical glitch).
Period: 3 Month Follow-up
Arm/Group | SOLVE-IT | Waitlist Control
Started | 444 | 491
Completed | 294 | 334
Not Completed | 150 | 157
Not completed — Participant would not respond | 150 | 157
Period: 6 Month Follow-up
Arm/Group | SOLVE-IT | Waitlist Control
Started | 444 (Completion of 3 month follow-up was not required for 6-month eligibility.) | 491 (Completion of 3 month follow-up was not required for 6-month eligibility.)
Completed | 311 | 350
Not Completed | 133 | 141
Not completed — Participant would not respond | 133 | 141

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOLVE-IT | Waitlist Control | Total
Number analyzed (Participants) | 444 | 491 | 935
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 444 | 491 | 935
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (1.7) | 21.3 (1.8) | 21.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 444 | 491 | 935
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 338 | 349 | 687
  Latino/Hispanic | 55 | 76 | 131
  Black/African American | 51 | 66 | 117
Region of Enrollment [Number; unit: participants] — Young MSM were recruited nationally over the web from each of the 50 states in the United States
  participants
    United States | 444 | 491 | 935
Counts of unprotected anal intercourse (UAI) past 3 months [Mean (Standard Deviation); unit: counts] | 11.7 (12.5) | 12.5 (11.8) | 12.12 (12.14)
Level of shame [Mean (Standard Deviation); unit: units on a scale] — Measures of reported shame (items from an existing subscale of Watson and Clark's (1994) Positive and Negative Affect Schedule-- the subscale is designed to assess State Shame). Participants indicate to what extent they experienced emotions that were part of this sub scale, responding on a scale from 1 (very slightly or not at all) to 5(extremely). Values reported represent the mean value per participant on the State Shame subscale; values per participant on this subscale therefore ranged from 1 to 5. Higher scores represent a higher level of reported state shame.
  units on a scale | 1.7 (.77) | 1.7 (.82) | 1.7 (.80)

OUTCOME MEASURES:

1. Primary Outcome: Residualized Change in Counts of Unprotected Anal Intercourse at 3 Months
Description: Counts of unprotected anal intercourse (one each for insertive and receptive; UAI) in the past 3 months with a non-primary partner were reported by participants at baseline, and 3 month follow-up. Reports of insertive and receptive anal intercourse per time period were summed. Change in unprotected anal intercourse was calculated at 3 months using residualized change scores (regressing 3-month reported UAI (Y) on baseline UAI. Negative numbers reflect a reduction in UAI over time). Although raw counts of UAI are heavily tailed, residualized change scores yield a normal distribution.
Time Frame: Measured at baseline and 3 month follow-up
Population: In SOLVE-IT at 3 months, 10 multivariate outliers were excluded based on Mahalanobis distance; in Wait-list Control 12 multivariate outliers were excluded.
Measure: Mean (Standard Deviation); unit: Res. Change in Counts of UAI at 3 months
Groups:
- Waitlist Control: After a 3-month waitlist period, participants will receive the intervention, SOLVE-IT, a video game designed to optimize self-regulation reduce shame, and reduce risky sexual choices for YMSM.
  SOLVE-IT: SOLVE-IT, a video game using computer-generated virtual agents, is the next generation of interactive media aimed at reducing risky sex among young MSM. Participants will interact in a virtual environment that focuses upon HIV prevention in a dating context.
Arm/Group | SOLVE-IT | Waitlist Control
Number analyzed (Participants) | 284 | 322
Res. Change in Counts of UAI at 3 months | .10 (6.67) | -.09 (9.95)

2. Primary Outcome: Residualized Change in Counts of Unprotected Anal Intercourse at 6 Months
Description: Counts of unprotected anal intercourse (one each for insertive and receptive) in the past 3 months with a non-primary partner were reported by participants at baseline, and 6 month follow-up. Reports of insertive and receptive anal intercourse per time period were summed. Change in unprotected anal intercourse from baseline, was calculated at 6 months using residualized change scores (regressing 6-month reported UAI (Y) on baseline UAI. Negative numbers reflect a reduction in UAI over time). Raw counts of UAI are heavily tailed, but residualized change scores are normally distributed.
Time Frame: Measured at baseline and 6 month follow-up
Population: Here we use only complete data for a given analysis. Using Mahlolanobis distance critical values 11 participants in the SOLVE-IT group and 5 participants in the Waitlist Control were multivariate outliers.
Measure: Mean (Standard Deviation); unit: Change in Counts of UAI at 6 months
Groups:
- Waitlist Control: After a 6-month waitlist period, participants will receive the intervention, SOLVE-IT, a video game designed to optimize self-regulation reduce shame, and reduce risky sexual choices for YMSM.
  SOLVE-IT: SOLVE-IT, a video game using computer-generated virtual agents, is the next generation of interactive media aimed at reducing risky sex among young MSM. Participants will interact in a virtual environment that focuses upon HIV prevention in a dating context.
Arm/Group | SOLVE-IT | Waitlist Control
Number analyzed (Participants) | 300 | 345
Change in Counts of UAI at 6 months | -.48 (3.95) | .41 (4.68)
Statistical Analysis 1: Comparison: SOLVE-IT vs Waitlist Control; Test type: Superiority; p < .001, t-test, 2 sided

3. Secondary Outcome: Shame Residualized Change
Description: Measures of reported shame (five items from an existing subscale of Watson and Clark's (1994) Positive and Negative Affect Schedule- Expanded Form-- designed to assess State Shame): ashamed, blameworthy, angry at self, disgusted with self, dissatisfied with self. Participants indicate to what extent they experienced emotions that were part of this sub scale, responding on a scale from 1 (very slightly or not at all) to 5(extremely). Values reported represent the mean value per participant on the State Shame subscale; values per participant on this subscale therefore ranged from 1 to 5. Higher scores represent a higher level of reported state shame. Scores on this scale are heavily tailed. Therefore, we have consistently used residualized change scores: This is calculated from baseline to immediate post; negative numbers for residualized change mean reduced shame baseline to immediate post.
Time Frame: Measured at baseline and Immediate post
Population: At baseline 443 (of 444) SOLVE-IT and 491 WLC filled out the shame measure, but 7 per condition responded with "refuse to answer". A technical glitch post-game (that affected immediate post baseline measures only) resulted in 337 participants in SOLVE-IT but 482 WLC responding to immediate post.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOLVE-IT | Waitlist Control
Number analyzed (Participants) | 337 | 482
score on a scale | -.13 (.65) | .09 (.03)

ADVERSE EVENTS:
Time Frame: 6 months per participant in the main study
Description: An approved data and safety monitoring plan stated that if three or more adverse events (e.g., distress, upset) occurred in a single arm, the trial would be stopped and evaluated. An adverse event form was developed for this purpose. Staff was trained to notify the Co-PI (and he the PI) immediately if one occurred (no adverse event occurred).
Arm/Group | SOLVE-IT | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/444 | 0/491
Other Adverse Events (participants affected / at risk) | 0/444 | 0/491

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No